CLINICAL TRIAL: NCT04534881
Title: Effect of Progesterone on Testosterone Concentrations and Breast Development in Transwomen
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of recruitment
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Sandeep Singh Dhindsa, M.D., F.A.C.E, Professor of Medicine, St. Louis University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 31144
Record Dates: First submitted 2020-08-17; First posted 2020-09-01 (Actual); Results first posted 2024-03-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-02

CONDITIONS: Transgender Persons
Keywords: Testosterone, breast
MeSH Terms: interventions — Progesterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- progesterone (Active Comparator): subjects on active drug (progesterone)
  Interventions: Drug: Progesterone 200 MG
- placebo (Placebo Comparator): subjects on placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Progesterone 200 MG — Subjects will be randomized to receive generic micronized progesterone 200 mg or placebo tablets, to be taken at bedtime daily.
  Arms: progesterone
Drug: Placebo — Subjects will be randomized to receive generic micronized progesterone 200 mg or placebo tablets, to be taken at bedtime daily.
  Arms: placebo

SUMMARY:
* Purpose. The purpose of this research is study the effect of progesterone therapy on testosterone levels in transwomen who are currently on gender affirming treatment with estradiol.
* Duration. It is expected that participation will last for 6 months (24 weeks).
* Study Procedures. Participants will be asked to sign an informed consent, complete a medical history, have a physical exam conducted, have a fasting blood sample taken and asked to take a study drug once daily.
* Risks. Some of the foreseeable risks or discomforts include temporary discomfort, bleeding, bruising and/or swelling in the arm from blood draw. There are no known direct risks with the use of Progesterone in Transwomen for gender affirming therapy.
* Benefits. Some of the possible benefits that may be expected include increase in fat mass, increase in breast size/fullness, decrease in masculine hair patterns.

DETAILED DESCRIPTION:
The number of individuals with gender incongruence who present to their physician for hormone therapy has increased manifold in the last decade. Testosterone therapy in transgender men (also known as female-to-male transgender or transmen) and estrogen therapy in transgender women (also known as male-to-female transgender or transwomen) respectively is the mainstay of hormone regimen.Transwomen, who are genetically men, receive estradiol replacement with the aim of suppressing serum testosterone and achieving serum estradiol concentrations that mimic the serum concentrations of biological women. This leads to an increase in fat mass, breast growth and decreases in lean mass and masculine pattern hair. However, the results of these changes are often less than satisfactory and additional therapy is required.

Breast development is a major concern for transgender females. There is a great deal of variability among individuals, as evidenced during pubertal development.Transgender women do not achieve the same level of breast development as cisgender women do after puberty. Typically, transgender women plateau at Tanner stage III and half of the transgender women have a AAA cup size or less.Investigators plan to conduct a randomized, placebo controlled double blind study evaluating the effect of adding progesterone for 6 months to transwomen who are being treated with estradiol. The hypothesis is that progesterone will decrease serum testosterone concentrations as compared to placebo and increase breast size. Investigators will also assess its role in mood, sleep, scalp hair and androgenic hair growth.

ELIGIBILITY:
Inclusion Criteria:

* Transwomen, currently on treatment with estradiol therapy for at least 6 months (as their standard of care gender affirming therapy)
* Has achieved serum estradiol >100 pg/ml at least once, based on clinical labs in past.

Exclusion Criteria:

1. Treatment with progesterone in the last 2 months
2. HIV
3. Planning to go for breast enhancement or gender reassignment surgery in the next 6 months
4. Known history of peanut allergy (because the study drug contains peanut oil)
5. Active deep vein thrombosis, pulmonary embolism or history of these conditions
6. Active arterial thromboembolic disease or history of these conditions
7. Active cardiovascular disorders or history of these conditions (e.g. myocardial infarction, uncontrolled hypertension >150/90 mmHg)
8. Known, suspected, or history of breast cancer
9. Known liver dysfunction or disease
10. Known or history of gallbladder disease. This does not apply to subjects who have undergone cholecystectomy
11. Known or history of hypertriglyceridemia (>400 mg/dl)

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Transwomen
Enrollment: 5 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2023-01-18 (Actual); Study Completion 2023-01-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandeep Singh Dhindsa Dhindsa, MD, Principal Investigator — St. Louis University
Locations (1):
- Saint Louis University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Progesterone: subjects on active drug (progesterone)
  Progesterone 200 MG: Subjects will be randomized to receive generic micronized progesterone 200 mg tablets, to be taken at bedtime daily.
- Placebo: subjects on placebo
  Placebo: Subjects will be randomized to receive placebo tablets, to be taken at bedtime daily.
Period: Overall Study
Arm/Group | Progesterone | Placebo
Started | 3 | 2
Completed | 3 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Progesterone | Placebo | Total
Number analyzed (Participants) | 3 | 2 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.7 (2.5) | 24.5 (0.7) | 28.8 (4.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 3 | 2 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 2 | 5
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Efficacy: Testosterone
Description: Change from baseline till 24 weeks in serum testosterone concentrations between progesterone and placebo groups. Calculated as testosterone levels at 24 weeks minus baseline
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Progesterone | Placebo
Number analyzed (Participants) | 3 | 2
ng/dL | 1.5 (4) | -6.4 (0)

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Progesterone | Placebo
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/2
Other Adverse Events (participants affected / at risk) | 0/3 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-13): https://cdn.clinicaltrials.gov/large-docs/81/NCT04534881/Prot_SAP_001.pdf